CLINICAL TRIAL: NCT02195141
Title: Randomized Phase II Tiral of Using SIB-IMRT in Preoperative Radiotherapy for Locally Advanced Rectum Cancer
Brief Title: Trial of Using SIB-IMRT in Preoperative Radiotherapy for Locally Advanced Rectum Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hua Ren, Attending physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC2014-ST02
Record Dates: First submitted 2014-07-11; First posted 2014-07-21 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Rectal Cancer
Keywords: Preoperative Chemoradiotherapy; Locally Advanced Rectal Cancer; boost; IMRT
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional fraction (Active Comparator): Radiotherapy (25x 2 Gy) + capecitabine 825mg/m2 p.o. twice daily
  Interventions: Radiation: conventional fraction
- SIB (Experimental): Concomitant chemoradiotherapy Radiotherapy with boost Radiotherapy (25 x 2 Gy), with a simultaneous integrated boost up to 56 Gy on the primary tumor capecitabine 825mg/m2 p.o. twice daily
  Interventions: Radiation: SIB

INTERVENTIONS:
Radiation: conventional fraction — capecitabine 825mg/m2 p.o. twice daily Radiotherapy 50Gy/25f
  Arms: conventional fraction
Radiation: SIB — Concomitant chemoradiotherapy Radiotherapy with boost Radiotherapy (25 x 2 Gy), with a simultaneous integrated boost up to 56 Gy on the primary tumor capecitabine 825mg/m2 p.o. twice daily
  Arms: SIB

SUMMARY:
Pathological complete response, (pCR) correlates with a favorable overall prognosis in locally advanced rectal cancer patients underwent preoperative chemoradiation, so obtaining a pCR might be beneficial. The aim of the study is to investigate safety and efficacy of preoperative SIB-IMRT(56Gy) combine with capecitabine. primary endpoint is pathological complete remission rate.

ELIGIBILITY:
Inclusion Criteria:

* histopathologically confirmed rectal adenocarcinoma with an inferior border within 15 cm of the anal verge
* the tumor has to have evidence of T3 or T4 disease on Magnetic Resonance Imaging (MRI) or endoluminal ultrasound

Exclusion Criteria:

* metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status > 3
* patients not deemed fit for radiotherapy, capecitabine or surgery
* pregnant or lactating patients
* women with child bearing potential who lack effective contraception
* patients below 18 years old

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
• Pathological complete remission rate (pCR) | after pathological examination of surgical speciments (6-8 weeks after chemoradiation)

SECONDARY OUTCOMES:
Number of participants with adverse events (according to the National Cancer Institute (NCI) - Common Terminology Criteria for Adverse Events v3.0 (CTCAE) | during preoperative treatment and after surgery for 5 years
  Acute toxicities will be assessed every week during chemoradiation period , one week before surgery(6 weeks after chemoradiation) and every 3 months after surgery for 2 years.Late toxicities will be assessed every 6 months from the 3rd year for 3 years.Adverse eventswill be evaluated according to the National Cancer Institute (NCI) - Common Terminology Criteria for Adverse Events v3.0 (CTCAE)

OTHER OUTCOMES:
• Disease-free survival | 3 year afte concurrent chemoradiation
  Followup will be done every 3 months in first 2 years, and every 6 months after 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Jin, proffessor, Study Chair — Dept of Radiation oncology, Cancer hospital, CAMS
Locations (1):
- Cancer Hospital, CAMS, Beijing, China